CLINICAL TRIAL: NCT03718572
Title: Evaluation Of Preoperative Scoring Method For Peridiction Of Difficult Laparoscopic Cholecystectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, AbdElRhman Mohamed Ahmed, Resident, Assiut University
Other Study IDs: AssiutU1001
Record Dates: First submitted 2018-10-23; First posted 2018-10-24 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Evaluation Studies
MeSH Terms: interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Scoring factors
  Interventions: Procedure: Laparoscopic cholecystectomy
- Difficulty criteria
  Interventions: Procedure: Laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: Laparoscopic cholecystectomy — Surgical removal of Gall bladder using laparoscopy

SUMMARY:
Registering and observing clinical and radiological data of patients undergoing laparoscopic cholecystectomy, then formulating these data aiming to find helpful scoring system to predict difficulty of laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Patients with symptomatic chronic calculous cholecystitis based on clinical and radiological correlation undergoing elective laparoscopic cholecystectomy at Assiut University hospitals will be included for the study of 30 patients will operated by single experienced laparoscopic surgeon.The scores are given on history, clinical examination and radiological findings one day prior to surgery on admission.

ELIGIBILITY:
Inclusion Criteria:

* Adults male and female age of or above 18 years
* Symptomatic chronic calculous cholecystitis
* Ultrasound confirmed Gall bladder stones

Exclusion Criteria:

* Complicated chronic calculous cholecystitis
* Malignant Gall bladder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults male and female age of or above 18 years
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of preoperative scoring method for prediction of difficult laparoscopic cholecystectomy | 6 monthes
  Validation of sensitivity and specificity of Scoring system to predict difficulty of laparoscopic cholecystectomy

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes